CLINICAL TRIAL: NCT01105884
Title: Clinical and Cost Effectiveness of Different Dressing Materials in Diabetic Foot Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to administrative reason
Sponsor: M.V. Hospital for Diabetes (Other)
Responsible Party: Principal Investigator, Vijay Viswanathan, MANAGING DIRECTOR, M.V. Hospital for Diabetes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDS01
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Foot Ulcers
Keywords: Wound healing, type 2 diabetes, diabetic foot ulcers, different dressings
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2 | interventions — Saline Solution; Colloids; Hydrogels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Active Comparator)
  Interventions: Procedure: Normal Saline
- Group 2 (Active Comparator)
  Interventions: Procedure: Biatin Ag (Foam)
- Group 3 (Active Comparator)
  Interventions: Procedure: Hydrocolloid
- Group 4 (Active Comparator)
  Interventions: Procedure: Hydrogel
- Group 5 (Active Comparator)
  Interventions: Procedure: Ceredak

INTERVENTIONS:
Procedure: Normal Saline — All the subjects in Group 1 will be treated with Normal Saline for healing of their diabetic foot ulcer
  Arms: Group 1
Procedure: Biatin Ag (Foam) — All the subjects will be treated with Biatin Ag (Foam)
  Other Names: Coloplast
  Arms: Group 2
Procedure: Hydrocolloid — All the subjects in this group will be treated with Hydrocolloid
  Other Names: Coloplast
  Arms: Group 3
Procedure: Hydrogel — All the subjects in this group will be treated with Hydrogel
  Other Names: Coloplast - Purilon Gel
  Arms: Group 4
Procedure: Ceredak — All the subjects in this group will be treated with Micro-porous Ceramic Wound Dressing
  Arms: Group 5

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of different commonly used dressings for treating diabetic foot ulcers. It is a prospective study recruiting 50 type 2 diabetic patients with diabetic foot ulcers (2-50cm2). All the patients will give written informed consent prior to getting enrolled in the study. All the patients will be randomly assigned to one of the five groups of the study namely, saline (control),Biatin Ag (Foam), Hydrocolloid, Hydrogel and Ceredak. Follow up of the patients will be done until the complete healing of the wound takes place. All procedures of dressing will be done by an authorized and certified Podiatric Surgeon of the Institution. Details on the cost incurred and days required for the wound to completely heal will be recorded for all the patients.

This study will provide the efficacy of all the dressings used for treating diabetic foot ulcers and also the cost of each dressing. This will help the surgeons for managing the diabetic foot ulcers in a better and cost effective way, which in turn will reduce the burden of patients both physically and financially.

DETAILED DESCRIPTION:
This prospective study aims at determining the efficacy and safety of different dressings available for treating diabetic foot ulcers. Study has been approved by the Institutional Ethics Committee before starting. Informed consent will be obtained from all the study subjects. A total of 50 subjects will be recruited. Study subjects will be divided in five groups of 10 subjects in each group.All the subjects will be randomly assigned to one of the study groups namely; Group 1 will the subjects randomized on Normal Saline (Control) and group 2 will be the subjects randomized on Biatin Ag (Foam) dressing; Group 3 will be Hydrocolloid, group 4 will be Hydrogel and Group 5 will be Ceredak. Lab investigations involving glycemic status (HbA1c), lipid profile, renal function test, liver function test will be done using standard enzymatic procedures. Wound size, colony count and microflora of the wound will be captured for all the study subjects. Photographs of the wound will be taken at every follow up visit until the wound is healed. Serum and tissue sample will be collected for the estimation of pronounced markers like MMP 2 and MMP 9. MMP 2 will be estimated using ELISA procedure (using standard enzymatic assay kit) and MMP 9 will be estimated using western blot technique. Histopathology of collagen will be seen using Van Gieson's stain. Immunohistochemistry will be done for determining collagen IV (marker for basement membrane thickening) to prove the evident wound healing at a defined point of time. H&E sections will be taken for determining the inflammation histochemically. All the study subjects will be followed till the wound healing process is complete. Tissue and serum samples will be collected for the above mentioned parameters on pre application day, after 1st and 4th week of the dressing application. A total of 3 visits will be performed for all the study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with foot ulcers
* Patients with or without PVD
* Size of the ulcer: 2-50 cm2
* Age 30-75 years (both gender)

Exclusion Criteria:

* Patient having severe infection
* Size of the foot ulcer > 50cm2
* Patients not willing to give written informed consent
* Patient with psychological disorder
* Patients with severe renal impairment or visual deformity
* Patients above the age of 75 years

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
complete healing of the wound | 1 months from the date of application

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Viswanathan, Dr, Principal Investigator — DRC; Rajesh Kesavan, Dr., Study Director — DRC
Locations (1):
- Diabetes Research Centre, Chennai, Tamil Nadu, India